CLINICAL TRIAL: NCT02438852
Title: Efficacy of Continuous Infusion of Local Anesthesia After Radical Cystectomy: A Randomized, Double Blind, Placebo Controlled Study
Brief Title: Continuous Infusion of Ropivacaine Hydrochloride in Reducing Pain After Surgery in Patients With Bladder Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4B-14-4; NCI-2015-00279 (Other: CTRP (Clinical Trial Reporting Program)); 4B-14-4 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Bladder Carcinoma; Post-operative Pain
MeSH Terms: conditions — Urinary Bladder Neoplasms; Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (ropivacaine hydrochloride) (Experimental): Patients receive ropivacaine hydrochloride IV continuously over 72 hours after radical cystectomy.
  Interventions: Other: Questionnaire Administration; Drug: Ropivacaine Hydrochloride
- Arm II (placebo) (Placebo Comparator): Patients receive normal saline (placebo) IV continuously over 72 hours after radical cystectomy.
  Interventions: Other: Placebo; Other: Questionnaire Administration

INTERVENTIONS:
Other: Placebo — Given IV
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Other: Questionnaire Administration — Ancillary studies
Drug: Ropivacaine Hydrochloride — Given IV
  Other Names: Naropin; Ropivacaine Hydrochloride Monohydrate
  Arms: Arm I (ropivacaine hydrochloride)

SUMMARY:
This randomized phase IV trial studies how well the continuous infusion of ropivacaine hydrochloride works in reducing pain after surgery in patients with bladder cancer. Ropivacaine hydrochloride is an anesthetic drug used to decrease pain by numbing an area of the body without putting the patient to sleep. Continuous infusion of ropivacaine hydrochloride may reduce pain and improve the quality of life for patients after bladder surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if continuous infusion of local anesthesia (CILA) decreases post-operative pain after radical cystectomy (RC).

II. To determine if CILA reduces narcotic requirements after RC.

SECONDARY OBJECTIVES:

I. To determine if CILA decreases length-of-stay after RC. II. To determine if CILA improves patients satisfaction with post-operative pain control after RC.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive ropivacaine hydrochloride intravenously (IV) continuously over 72 hours after radical cystectomy.

ARM II: Patients receive normal saline (placebo) IV continuously over 72 hours after radical cystectomy.

After completion of study, patients are followed up within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective open radical cystectomy
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Allergy or adverse reaction to ropivacaine (ropivacaine hydrochloride) or any amide type of local anesthesia
* Allergy or adverse reaction to local anesthesia catheter
* Additional surgery at the same time as RC (e.g. nephroureterectomy)
* Coagulopathy
* Thrombocytopenia
* Local or systemic infection
* Pregnancy
* Chronic hepatic disease
* Use of type III antiarrhythmics (e.g. amiodarone)
* History of chronic pain and/or daily opioid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-25 (Estimated); Primary Completion 2021-02-25 (Estimated); Study Completion 2022-02-25 (Estimated)

PRIMARY OUTCOMES:
Narcotic requirement | Up to 72 hours after surgery
  Total narcotic dose after surgery until 72 hours will be analyzed as continuous variables and will be compared with the one sided t-test in an intention-to-treat manner.

SECONDARY OUTCOMES:
Length of hospitalization | Up to 30 days after surgery
  The length of hospitalization will be analyzed as continuous variables and will be compared with the one sided t-test in an intention-to-treat manner.

CONTACTS AND LOCATIONS:
Overall Officials: Siamak Daneshmand, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States